CLINICAL TRIAL: NCT03954301
Title: Anthropometric and Biomechanical Variables Causing Foot Deformities in Young Individuals, Using the Hierarchical Cluster Method
Brief Title: Using the Hierarchical Cluster Method for Foot Deformities
Acronym: Cluster
Status: Completed | Type: Observational
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Başar Öztürk, Assistant Professor, Biruni University
Other Study IDs: BiruniUni
Record Dates: First submitted 2019-05-14; First posted 2019-05-17 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Foot Deformities
Keywords: Foot deformities; Cluster method; Kinematic analysis
MeSH Terms: conditions — Foot Deformities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Anthropometric measures — Q, valgity angle, subtalar joint, medial longitudinal arch and hallux valgus angles were measured with a goniometer. The height from the ground of the navicula was calculated by caliper, using the Navicular drop test. Metatarsal width was also calculated with this device. Medial longitudinal arch angle, metatarsal width and nacivular drop tests were performed under weight-bearing and non-weight-bearing conditions.
  Other Names: Kinematic analysis

SUMMARY:
The aim of this study is to analyze all of the variables with a Hierarchical Cluster Analysis of Multivariate Statistical Methods to obtain more sensitive results, and also to add a new dimension to the hypothesis included in the study.

DETAILED DESCRIPTION:
Aim and Introduction: Due to individual anthropometric differences, there are many different types of foot posture Foot posture variations affect lower extremity structure, alignment and biomechanical characteristics. Particularly in younger people, performing critical biomechanical measurements in the lower extremity and foot is extremely important to the detection of, and early intervention in, orthopedic problems that these individuals will encounter in their later life. In the literature, attempts at analysis of the evaluations realized so far have been made by univariate analysis. Considering the relationship between variation and variables, these methods result in loss of information. The aim of this study is to analyze all of the variables with a Hierarchical Cluster Analysis of Multivariate Statistical Methods to obtain more sensitive results, and also to add a new dimension to the hypothesis included in the study.

Methods: The study is carried out on 2nd and 3rd year university students in the physiotherapy and rehabilitation department taking a kinesiology course. The analyses are performed at the Biruni University Physiotherapy and Rehabilitation laboratory. Patients with musculoskeletal system pathomechanics which could prevent standing and walking are not included in the study. After demographic characteristics are recorded, Q, valgity angle, subtalar joint, medial longitudinal arch and hallux valgus angles are measured with a goniometer. The height from the ground of the navicula are calculated by caliper, using the Navicular drop test. Metatarsal width are also calculated with this device. Medial longitudinal arch angle, metatarsal width and nacivular drop tests are performed under weight-bearing and non-weight-bearing conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy university students.
* Must be able to walk independently.

Exclusion Criteria:

* Students with chronic sprains.
* Students who had undergone lower extremity surgery within the last year.
* Students who use assistive walking devices.

Ages: 18 Years to 24 Years | Sex: All
Age Groups: Adult
Study Population: University students
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Navicular drop test | 2 weeks.
  The height of navicula will be measured in weight-bearing and non-weight bearing conditions in millimeters.
Metatarsal width | 2 weeks.
  The width of metatarsal zone will be measured in weight-bearing and non-weight bearing conditions in millimeters.
Subtalar angle | 2 weeks.
  The angle between calcaneus and Achilleus tendon will be measured with goniometer in standing position and the degree will be calculated.
Hallux valgus angle | 2 weeks.
  The angle between 1st metatars and hallux will be measured with goniometer and the degree will be calculated.

SECONDARY OUTCOMES:
Q angle | 2 weeks.
  The angle of quadriceps femoris muscle will be measured with goniometer in supine position and the degree will be assessed.
Medial longitudinal arch angle | 2 weeks.
  The angle between 1st metatarsophalangeal joint, navicula and medial malleol will be measured and the degree will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Başar Öztürk, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No